CLINICAL TRIAL: NCT02046265
Title: Step up to Prevention : A Nurse Practitioner Guided Cervical Cancer Prevention Intervention
Brief Title: Clinic-based Intervention to Promote Cervical Cancer Prevention Behaviors
Acronym: StepUp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: StepUpToPrevention
Record Dates: First submitted 2014-01-14; First posted 2014-01-27 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-06

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Step Up to Prevention: knowledge (Experimental): Participant receives an individual computer-delivered information session and participant is offered the HPV vaccine only by their nurse practitioner in clinic.
  Interventions: Behavioral: Step Up to Prevention: knowledge
- Step Up to Prevention:belief (Experimental): Participant receives a one-on-one tailored educational session with a trained study team member and participant is offered the HPV vaccine only by their nurse practitioner in clinic.
  Interventions: Behavioral: Step Up to Prevention:belief
- Step up to Prevention (Experimental): Participant receives both the knowledge session and the tailored belief sessions and the participant is offered the HPV vaccine only by their nurse practitioner in clinic. This combined intervention is call Step Up to Prevention.
  Interventions: Behavioral: Step Up to Prevention
- Offered HPV vaccine only (Active Comparator): Participant is offered the HPV vaccine only by their nurse practitioner in clinic.
  Interventions: Behavioral: Offered HPV vaccine only

INTERVENTIONS:
Behavioral: Step Up to Prevention — Participant receives a one-on-one tailored educational session with a trained study team member and participant is offered the HPV vaccine only by their nurse practitioner in clinic.
  Arms: Step up to Prevention
Behavioral: Step Up to Prevention: knowledge — Participant receives an individual computer-delivered information session and participant is offered the HPV vaccine only by their nurse practitioner in clinic.
  Arms: Step Up to Prevention: knowledge
Behavioral: Step Up to Prevention:belief — Participant receives a one-on-one tailored educational session with a trained study team member and participant is offered the HPV vaccine only by their nurse practitioner in clinic.
  Arms: Step Up to Prevention:belief
Behavioral: Offered HPV vaccine only — Participant is offered the HPV vaccine only by their nurse practitioner in clinic.
  Arms: Offered HPV vaccine only

SUMMARY:
The project is a clinical behavioral research project based at University of Pennsylvania. The goal of this research is to design a brief clinic-based, Nurse Practitioner-guided, and theory-based health promotion intervention to enhance cervical cancer prevention among young women ages 18-26 living in economically disadvantaged urban communities. The investigators will evaluate the intervention for feasibility, acceptability and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-26 years
* Not yet received the HPV vaccine
* Speak, read, and understand 5th grade level of English;
* Had vaginal sex with a male partner in the past 2 months.

Exclusion Criteria:

• Currently pregnant and/or plan to be pregnant in next 6 months

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Teitelman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Outpatient Ob/GYN clinic, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 sites, both with federally-supported family planning programs.
Pre-assignment Details: All participants completed a baseline survey prior to randomization.
Period: Overall Study
Arm/Group | Step Up to Prevention: Knowledge | Step Up to Prevention:Belief | Step up to Prevention | Offered HPV Vaccine Only
Started | 17 | 17 | 12 | 14
Completed | 16 | 15 | 10 | 12
Not Completed | 1 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Step Up to Prevention: Knowledge | Step Up to Prevention:Belief | Step up to Prevention | Offered HPV Vaccine Only | Total
Number analyzed (Participants) | 17 | 17 | 12 | 14 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.06 (2.14) | 21.56 (2.00) | 21.75 (2.59) | 20.77 (1.80) | 21.54 (2.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 12 | 14 | 60
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 7 | 6 | 34
  White | 5 | 5 | 2 | 5 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 12 | 14 | 60

OUTCOME MEASURES:

1. Primary Outcome: Human Papilloma Virus (HPV) Vaccine #1 Acceptance
Time Frame: For each participant, at end of first study visit. Will assess until all subjects enrolled in study.
Population: All participants in the analysis were eligible to recieve the HPV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Step Up to Prevention: Knowledge | Step Up to Prevention:Belief | Step up to Prevention | Offered HPV Vaccine Only
Number analyzed (Participants) | 16 | 15 | 10 | 12
Participants | 13 | 12 | 7 | 3

ADVERSE EVENTS:
Time Frame: 21 months
Arm/Group | Step Up to Prevention: Knowledge | Step Up to Prevention:Belief | Step up to Prevention | Offered HPV Vaccine Only
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No